CLINICAL TRIAL: NCT05207137
Title: [In Norwegian]: Samtale Med Fastlegen Som Tiltak for å øke Covid-19-vaksinedekningen
Brief Title: Conversation With Family Doctor to Increase COVID-19 Vaccine Uptake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian Institute of Public Health (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Cristin-ID: 2526531
Record Dates: First submitted 2021-12-08; First posted 2022-01-26 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2022-01

CONDITIONS: COVID-19
Keywords: Health services research; Quality improvement
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Telephone call from family physician (Experimental): Individuals allocated to the experimental arm will receive a phone call from the their family physician, where they are offered the opportunity to raise questions they might have about the COVID-19 vaccine.
  Interventions: Behavioral: Telephone call about vaccination
- Usual care (No Intervention)

INTERVENTIONS:
Behavioral: Telephone call about vaccination — Participants receive phone call from their family physician, where they are invited to ask questions about the COVID-19 vaccine.
  Arms: Telephone call from family physician

SUMMARY:
The investigators will randomise individuals from family doctors' lists of patients that are at risk of severe Coronavirus Disease 2019 (COVID-19), and that are not registered as having taken the vaccine against the disease. The patients will be randomised to receiving a phone call from their family physician where the participants are given the opportunity to raise questions they might have around vaccination. The investigators will assess whether this has an impact on vaccine uptake.

ELIGIBILITY:
Inclusion Criteria:

* Belonging to group at risk of severe COVID-19

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 654 (Actual)
Dates: Start 2021-12-03 (Actual); Primary Completion 2022-04-28 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Vaccination status (COVID-19) | 3-6 weeks after inclusion
  Change in proportion of participants who are registered in the national vaccination registry, as having received at least one dose of a COVID-19 vaccine.

CONTACTS AND LOCATIONS:
Overall Officials: Atle Fretheim, PhD, Study Director — Norwegian Institute of Public Health
Locations (1):
- Bolteløkka legesenter, Oslo, Norway

REFERENCES:
- [Background] Tuv M, Elgersma IH, Furuseth E, Holst C, Helleve A, Fretheim A. GP phone calls to improve COVID-19 vaccine uptake among patients at increased risk of severe COVID-19: a randomised trial. BJGP Open. 2023 Jun 27;7(2):BJGPO.2022.0175. doi: 10.3399/BJGPO.2022.0175. Print 2023 Jun. PMID 36754551
- See also: Main study report — https://bjgpopen.org/content/early/2023/02/06/BJGPO.2022.0175